CLINICAL TRIAL: NCT01535079
Title: Analgesic Profile of 3 New Ibuprofen Lozenges (V0498TA01A 15 mg, 25 mg, 35 mg) After Single Administration in Acute Sore Throat Pain
Brief Title: Acute Sore Throat Pain Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: V00498 TA 2 01; 2011-005848-10 (EudraCT Number)
Record Dates: First submitted 2012-02-10; First posted 2012-02-17 (Estimated); Last update posted 2012-11-12 (Estimated); Status verified 2012-10

CONDITIONS: Acute Sore Throat Pain
Keywords: sore throat pain; tonsillopharyngitis; upper respiratory tract infection
MeSH Terms: conditions — Respiratory Tract Infections | interventions — Ibuprofen; Flurbiprofen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (5):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- V0498TA01A 15 mg (Experimental)
  Interventions: Drug: Ibuprofen 15 mg
- V0498TA01A 25 mg (Experimental)
  Interventions: Drug: Ibuprofen 25 mg
- V0498TA01A 35 mg (Experimental)
  Interventions: Drug: Ibuprofen 35 mg
- Strefen (Other): Positive control
  Interventions: Drug: Strefen

INTERVENTIONS:
Drug: Placebo — Single administration
  Arms: Placebo
Drug: Ibuprofen 35 mg — Single administration
  Arms: V0498TA01A 35 mg
Drug: Ibuprofen 25 mg — Single administration
  Arms: V0498TA01A 25 mg
Drug: Ibuprofen 15 mg — Single administration
  Arms: V0498TA01A 15 mg
Drug: Strefen — Single administration
  Arms: Strefen

SUMMARY:
"Sore throat is one of the most common complaints encountered in clinical practice. And in 65% of cases, the infection is thought to be viral in nature.

The aim of this study is to evaluate the analgesic profile of 3 Ibuprofen lozenges after single administration in acute sore throat pain."

ELIGIBILITY:
Inclusion Criteria:

* male or female patients 18 years and older
* patients with a sore throat associated or not with an Upper Respiratory Tract Infection ≥ 24 hours and ≤ 5 days duration, in the absence of Streptococcus group A

Exclusion Criteria:

* patients with hypersensitivity to Ibuprofen or other NSAIDs or the excipients.
* patients having used analgesics or antiseptics or any topical throat treatment or any local medication containing a local oral anaesthetic within 6 hours before study entry and who use analgesics more than ≥ 3 times per week.
* patients having used any anti inflammatory treatment or any long-acting or slow release analgesics within 12 hours before study entry
* patients having taken antibiotics within 14 days before study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2012-02; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline of Sore Throat Pain Intensity Scale | 60 minutes

SECONDARY OUTCOMES:
Change from baseline of Sore Throat Pain relief Scale | up to 360 minutes
Change of Sore Throat Pain Intensity Scales | up to 360 minutes
Local tolerability examination | Baseline (before drug intake) and 360 minutes
  Mouth examination including extent of erythema, edema, petechial hemorrhages, ulceration (4 point scale : none, mild, moderate and severe).
General tolerability (reported adverse events) | Baseline (before drug intake) and 360 minutes

CONTACTS AND LOCATIONS:
Locations (4):
- France (2):
  - Eurofins Optimed, Gières
  - Eurofins Optimed Lyon, Pierre-Bénite
- Erfurt, Germany
- Cardiff, United Kingdom